CLINICAL TRIAL: NCT06020378
Title: Hydroxychloroquine Treatment During Pregnancy is Associated With Lower Risk of Preeclampsia in Patients With Recurrent Spontaneous Abortion of Unknown Aetiology
Brief Title: Hydroxychloroquine May be Beneficial for Preeclampsia
Status: Active, not recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2022-0186
Record Dates: First submitted 2023-08-07; First posted 2023-08-31 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Hydroxychloroquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hydroxychloroquine treatment group: The Hydroxychloroquine treatment group was defined as having exposure to Hydroxychloroquine during pregnancy.
  Interventions: Drug: Hydroxychloroquine
- Hydroxychloroquine nontreatment group: The Hydroxychloroquine nontreatment group was defined as having no exposure to Hydroxychloroquine during pregnancy.

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine was administered during pregnancy
  Other Names: Plaquenil
  Groups: Hydroxychloroquine treatment group

SUMMARY:
The purpose of this research is to investigate the impact of hydroxychloroquine on the incidence of hypertensive pregnancy disorders in women with a history of recurrent spontaneous abortion (RSA).

DETAILED DESCRIPTION:
Preeclampsia affects about 3-5% of all pregnancies and is estimated to cause at least 42 000 maternal deaths annually, remaining an important cause of death and complications for the mother and baby. However, no treatment yet has been found that affects disease progression except for termination of pregnancy which may cause iatrogenic preterm labor. Therefore, keenly sought for approaches to improving clinical outcomes in pre-eclampsia would be needed.

Hydroxychloroquine (HCQ), an antimalarial drug, is commonly used in the treatment of pregnant women with RSA and has proven to be safe for both the mother and the fetus. Because of the antioxidant effect, anti-inflammatory effect, and vasculoprotective effect of HCQ, it has been thought to be beneficial in the prevention of preeclampsia.

Therefore, we conducted a retrospective cohort study to evaluate the impact of HCQ treatment on the prevention of preeclampsia in RSA pregnancies.

ELIGIBILITY:
Inclusion Criteria:

1. singleton pregnant women
2. with a history of two or more miscarriages

Exclusion Criteria:

1. indication to a treatment according to the severe cardiovascular, immune, respiratory, gastrointestinal/liver and biliary system, kidney and urinary system, nervous system, musculoskeletal system, psychiatric, infectious disease, malignancy,
2. major malformation of the fetus diagnosed at 11-13 weeks of gestation.
3. Known paternal, maternal, or embryo chromosome abnormality;
4. Abnormal uterine anatomy at hysterosalpingography/hysteroscopy or hydrosonography that might explain RM in the first trimester of pregnancy;
5. Maternal endocrine dysfunction: premature ovarian failure, hyperprolactinemia, corpus luteal insufficiency, untreated diabetes mellitus or untreated thyroid dysfunction.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women with RSA who delivered after 28 weeks from November 2016 to August 2022 at Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite morbidity | Gestational period
  Preeclampsia, gestational hypertension, preeclampsia superimposed upon chronic hypertension

SECONDARY OUTCOMES:
fetal growth restriction | 37 weeks of gestational age
  <10th percentile for gestational age
Preterm delivery | 37 weeks of gestational age
  Delivery before 37 weeks
Abruptio placenta | 37 weeks of gestational age
  The number of cases of abruptio placenta that appear in both groups at any given time during pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University School of Medicine，Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided